CLINICAL TRIAL: NCT01116583
Title: The Effect of Gabapentin on Thoracic Epidural Analgesia Following Thoracotomy - A Randomized, Double-blind, Placebo-controlled Trial
Brief Title: The Effect of Gabapentin on Thoracic Epidural Analgesia Following Thoracotomy
Acronym: GABATEA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital Skejby (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2007-002769-11
Record Dates: First submitted 2010-04-27; First posted 2010-05-05 (Estimated); Last update posted 2014-08-05 (Estimated); Status verified 2012-09

CONDITIONS: Pain, Postoperative
Keywords: Gabapentin; Thoracotomy; Pain, Postoperative; Analgesia; Recovery of Function; Quality of Life
MeSH Terms: conditions — Pain, Postoperative; Agnosia | interventions — Gabapentin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Gabapentin (Active Comparator): Gabapentin group
  Interventions: Drug: Gabapentin
- Placebo (Placebo Comparator): Placebo group
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Gabapentin — Preoperatively (2 hours before surgery): 4 gabapentin capsules each containing 300 mg gabapentin (total gabapentin dose 1200 mg)
  Postoperative day 1: gabapentin 300 mg x 2 (total gabapentin dose 600 mg)
  Postoperative day 2: gabapentin 300 mg x 3 (total gabapentin dose 900 mg)
  Postoperative day 3: gabapentin 300 mg x 4 (total gabapentin dose 1200 mg)
  Postoperative day 4: gabapentin 300 mg x 4 (total gabapentin dose 1200 mg)
  Postoperative day 5: gabapentin 300 mg x 4 (total gabapentin dose 1200 mg)
  Other Names: Gabapentin "Sandoz" 300 mg
  Arms: Gabapentin
Drug: Placebo — Preoperatively (2 hours before surgery): 4 placebo capsules
  Postoperative day 1: 1 placebo capsule x 2
  Postoperative day 2: 1 placebo capsule x 3
  Postoperative day 3: 1 placebo capsule x 4
  Postoperative day 4: 1 placebo capsule x 4
  Postoperative day 5: 1 placebo capsule x 4
  Arms: Placebo

SUMMARY:
The purpose of this trial is to investigate the effect of gabapentin on thoracic epidural analgesia following thoracotomy, including assessment of both analgesia, pain intensity, pain quality and whether or not gabapentin prevents the development of chronic pain conditions following thoracotomy.

The main hypothesis is that gabapentin reduces the proportion of patients who develop a persistent pain condition following thoracotomy from 50% to 20%.

Furthermore gabapentin is expected to reduce both pain intensity measured on a 11-point numerical rating scale, usage of epidural infusions of local and/or opioid analgesics, morbidity, hospital length of stay, consumption of opioid analgesics and analgesia-related side-effects.

In addition gabapentin is expected to improve postoperative recovery by means of postoperative lung function, walking ability, health related quality of life and patient satisfaction

ELIGIBILITY:
Inclusion Criteria:

* Elective lung resection via thoracotomy
* Age > 18 and < 80 years

Exclusion Criteria:

* Inability to answer the detailed questionnaires on pain and quality of life
* Psychiatric disease (ICD-10)
* Severe renal impairment (se-creatinin > 110 mmol/l)
* Known allergy to gabapentin, morphine, bupivacaine and / or ibuprofen
* Standard use of opioid analgesics
* Treatment with anticonvulsants or tricyclic antidepressants
* Use of antacids 24 hours before the intake of study medication
* Contraindicated placement of a thoracic epidural catheter
* Previous ipsilateral thoracotomy
* Presence of a chronic pain syndrome
* Acute pancreatitis
* A history of past or current alcohol and / or illegal substance abuse.
* A history of gastric or duodenal ulcer
* Gastrointestinal obstruction
* Pregnancy
* Participation in another intervention study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2011-05; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Persistent post surgical pain | 3 months after surgery
  Pain is assessed by means of the Brief Pain Inventory (BPI-SF) and The McGill Pain Questionnaire (SF-MPQ). Persistent postoperative pain is measured both on a 11-point numeric pain rating scale and on a 10 cm visual analog scale (VAS). A score >=3 is considered as moderate pain.
Acute postoperative pain | Within the first 5 postoperative days
  Acute postoperative pain is measured on a 11-point numeric rating scale both at rest and when coughing/sitting up. General pain intensity and specific (shoulder) pain intensity are measured. On postoperative day 4 pain is furthermore assessed by means of the Brief Pain Inventory (BPI-SF) and The McGill Pain Questionnaire (SF-MPQ). A score >=3 is considered as moderate pain.
Usage of epidural infusion of local and opioid analgesics (ml) | Within the first 5 postoperative days
Persistent post surgical pain | 6 months following surgery
  Pain is assessed by means of the Brief Pain Inventory (BPI-SF) and The McGill Pain Questionnaire (SF-MPQ). Persistent postoperative pain is measured both on a 11-point numeric pain rating scale and on a 10 cm visual analog scale (VAS). A score >=3 is considered as moderate pain.
Persistent post surgical pain | 12 months following surgery
  Pain is assessed by means of the Brief Pain Inventory (BPI-SF) and The McGill Pain Questionnaire (SF-MPQ). Persistent postoperative pain is measured both on a 11-point numeric pain rating scale and on a 10 cm visual analog scale (VAS). A score >=3 is considered as moderate pain.
Early postoperative pain | 14 days (+/-3 days) following discharge
  Early postoperative pain is measured on day 14 (+/-3 days) following discharge pain using the Brief Pain Inventory (BPI-SF) and The McGill Pain Questionnaire (SF-MPQ). A score >=3 is considered as moderate pain.

SECONDARY OUTCOMES:
Consumption of opioid analgesics | Within the first 5 postoperative days
Time to first request for additional analgesics | Within the first 5 postoperative days
Analgesia related side-effects | Within the first 5 postoperative days
  Evaluation of the presence and/or severity of confusion, hallucinations, nausea, vomiting, usage of antiemetic drugs, urinary retention, sedation, pruitus, headache, respiratory depression, motor blockade and dizziness
Convalescence of gastrointestinal function | Within the first 5 postoperative days
  Convalescence of gastrointestinal function (time to first defecation)
Health related quality of life | Day 14 (+/-3 days) following discharge
  Health related quality of life is measured with the EORCT QLQ-C30 and EORCT QLQ-LC13 questionnaires.
Patient satisfaction | Within the first 5 postoperative days
  Patient satisfaction is assesed with the EORCT-INPATSAT32 questionnaire
Intensity of preoperative anxiety | 2 hours after administration of the first dose of study medication
  Anxiety is measured on a 11-point numeric rating scale (NRS).
Convalescence of lung function (spirometry) | Within the first five postoperative days
  FVC, FEV-1 and PEF is measured.
Sleep quality | Within the first five postoperative days
  Sleep quality is measured on a 11-point numeric rating scale (NRS)
Walking distance (meters) | Postoperative day 3
  Ability to walk is measured by means of the 6-minutes walking test on postoperative day 3.
Fatigue | Within the first 5 postoperative days
  Fatigue is measured on a 4-point verbal rating scale (0=None, 1=Mild, 2=Moderate, 3=Severe).
Hospital length of stay (days) | At time of discharge
Health related quality of life | 3 months following surgery
  Health related quality of life is measured with the EORCT QLQ-C30 and EORCT QLQ-LC13 questionnaires.
Health related quality of life | 6 months following surgery
  Health related quality of life is measured with the EORCT QLQ-C30 and EORCT QLQ-LC13 questionnaires.
Health related quality of life | 12 months following surgery
  Health related quality of life is measured with the EORCT QLQ-C30 and EORCT QLQ-LC13 questionnaires.
Use of a vasopressor agent to correct hypotension | Within the first 5 days of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Hans K Pilegaard, MD, Chief Surgeon, Principal Investigator — Department of Cardiothoracic and Vascular Surgery, Aarhus University Hospital, Skejby, Denmark; Kasper Grosen, RN, MHScS, PhDS, Study Director — Department of Cardiothoracic and Vascular Surgery, Aarhus University Hospital, Skejby, Denmark; Vibeke Hjortdal, MD, Professor, DMSc, PhD, Study Chair — Department of Cardiothoracic and Vascular Surgery, Aarhus University Hospital, Skejby, Denmark; Mogens P Jensen, MD, Chief Physician, PhD, Study Chair — Department of Reumatology, Aarhus University Hospital, Aarhus Hospital, Denmark; Gerhard Linnemann, MD, Chief Physician, Study Chair — Department of Anaesthesiology and Intensive Care, Aarhus University Hospital, Skejby, Denmark; Vibeke Laursen, RN, Study Chair — Department of Cardiothoracic and Vascular Surgery, Aarhus University Hospital, Skejby, Denmark; Anette Hoejsgaard, MD, Study Chair — Department of Cardiothoracic and Vascular Surgery, Aarhus University Hospital
Locations (1):
- Department of Cardiothoracic and Vascular Surgery, Aarhus University Hospital, Skejby, Aarhus N, Denmark